CLINICAL TRIAL: NCT02815527
Title: Time to Protein Target, the 'HIGH WHEY' Study A Prospective Pilot Study
Brief Title: Time to Protein Target Using a High Whey Protein Enteral Nutrition in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, H.M. Oudemans-van Straaten, MD, PhD, Prof. Dr., Amsterdam UMC, location VUmc
Other Study IDs: 2015.560
Record Dates: First submitted 2016-05-09; First posted 2016-06-28 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Critically Ill
Keywords: enteral nutrition; intensive care unit; whey; protein; muscle mass; leucin; energy expenditure
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Fresubin Intensive: Adult critically ill non-septic ventilated patients admitted to the intensive care unit with an expected intensive care stay of four days or more.
  Interventions: Other: Fresubin intensive

INTERVENTIONS:
Other: Fresubin intensive — Enteral nutrition containing a high protein concentration

SUMMARY:
This study evaluates the feasibility of a high whey-protein enteral nutrition formula in 20 ventilated ICU patients. The primary endpoint of study is the feasibility to attain the individualized protein target (≥1.2 g/kg ideal body weight/day) 96-hours after ICU admission. Secondary endpoints include tolerance and efficacy in terms of the amino acid response in blood.

DETAILED DESCRIPTION:
In the present pilot study, the investigators will use a high whey-protein nutrition formula during the first four days of ICU admission. The reason for using a high protein nutrition is that the investigators previously found that an early high protein intake in non-septic non-overfed patients was associated with lower hospital mortality (Weijs PJM et. al., Critical Care 2014,18). Furthermore, during the first days of critical illness tolerance to full enteral nutrition is often diminished. The use of a high protein nutrition will facilitate an early high protein intake.

The whey protein is hydrolysed. Hydrolyzation of protein prevents coagulation and subsequent solidification in the digestive tract and therefore promotes efficient absorption of the protein. Of all nutrition proteins, whey protein has the largest leucin content. Leucin is crucial for muscle protein synthesis. (Meyer RF, et.al.: BMC Gastroenterol 2015, 15), (Marik PE: Ann Intensive Care 2015,5:51)

Our previous observational data also showed that early overfeeding was associated with higher mortality, while an intake of 80-100% of measured energy expenditure at day 4 of ICU admission was associated with lower mortality. (Weijs PJM et. al., Critical Care 2014, 18)

Therefore, the energy target during the first four days will be 90% of the measured Energy Expenditure (EE). To optimize energy intake, the investigators will measure EE by metabolic monitoring (Deltatrac®, Datex, Helsinki, Finland), If metabolic monitoring is not available, the investigators will assess EE from the ventilator derived VCO2 (8.19*VCO2). (Stapel S, et.al., Critical Care 2015,19:370)

ELIGIBILITY:
Inclusion Criteria:

* Admission to the intensive care unit
* Age >18 years
* Mechanical ventilation
* Expected intensive care stay of four days or longer

Exclusion Criteria:

* Contraindication for enteral nutrition (gut ischemia, obstruction or perforation)
* Expected intolerance for enteral nutrition (paralytic ileus)
* Inability to start enteral nutrition within 24-hours due to logistic reasons (i.e. surgery or other interventions)
* Short bowel syndrome
* Child C liver cirrhosis or acute liver failure
* Dialysis dependency
* Requiring other specific enteral nutrition for medical reason
* Extensive treatment limitations
* Written deferred patient or proxy consent is not obtained
* Participation in another intervention study
* Inability to measure energy expenditure (pulmonary air leakage)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ventilated critically ill patients in the ICU
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-03; Primary Completion 2017-06 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
The proportion of patients reaching the individualized protein target (≥1.2 g/kg ideal body weight/day) 96 hours after ICU admission | 96 hours
  Protein target

SECONDARY OUTCOMES:
Protein intake 48 hours and 96 hours after start (g/day) | 48 and 96 hours
  Protein intake
Number of patients with adverse events related to nutrition, as defined by: high gastric retention,abdominal distension, vomiting, diarrhea, need of prokinetics or duodenal tube | During 96 hours
  Gastro-intestinal tolerance
Plama leucine concentration (μmol/L) | 0, 48, and 96 hours
  Amino acid plasma concentration
Muscle mass (kg) | 48 and 96 hours
  Measured using bioimpedance analysis
Plasma urea concentration (mmol/l) | 48 and 96 hours
  Metabolic tolerance
Cumulative protein intake 96 hours after start of the study formula (grams) | 96 hours
  Cumulative protein intake
Time to protein target (protein intake ≥ 1.2 g/kg/day). | Up to 96 hours
  Time to target

CONTACTS AND LOCATIONS:
Overall Officials: Heleen M. Oudemans-van Straaten, MD. Prof., Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU Medical Center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meyer R, Foong RX, Thapar N, Kritas S, Shah N. Systematic review of the impact of feed protein type and degree of hydrolysis on gastric emptying in children. BMC Gastroenterol. 2015 Oct 15;15:137. doi: 10.1186/s12876-015-0369-0. PMID 26472544
- [Background] Marik PE. Feeding critically ill patients the right 'whey': thinking outside of the box. A personal view. Ann Intensive Care. 2015 Dec;5(1):51. doi: 10.1186/s13613-015-0051-2. Epub 2015 May 28. PMID 26055186
- [Background] Weijs PJ, Looijaard WG, Beishuizen A, Girbes AR, Oudemans-van Straaten HM. Early high protein intake is associated with low mortality and energy overfeeding with high mortality in non-septic mechanically ventilated critically ill patients. Crit Care. 2014 Dec 14;18(6):701. doi: 10.1186/s13054-014-0701-z. PMID 25499096
- [Background] Stapel SN, de Grooth HJ, Alimohamad H, Elbers PW, Girbes AR, Weijs PJ, Oudemans-van Straaten HM. Ventilator-derived carbon dioxide production to assess energy expenditure in critically ill patients: proof of concept. Crit Care. 2015 Oct 22;19:370. doi: 10.1186/s13054-015-1087-2. PMID 26494245